CLINICAL TRIAL: NCT06273111
Title: A Pilot Study Using Topical Statins to Treat Children With Infantile Hemangioma
Brief Title: Topical Simvastatin for Treating Infantile Hemangioma
Acronym: TSTIH
Status: Not yet recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Joyce Teng (Other)
Collaborators: Stanford University (Other)
Responsible Party: Sponsor-Investigator, Joyce Teng, Professor of Dermatology and Pediatric, Stanford University
Organization: Stanford University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 73840
Record Dates: First submitted 2024-02-15; First posted 2024-02-22 (Actual); Last update posted 2024-02-22 (Actual); Status verified 2024-02

CONDITIONS: Hemangioma Skin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- 5% simvastatin ointment (Experimental): Participants will be applied 5% simvastatin ointment on IH lesion
  Interventions: Drug: 5% simvastatin ointment

INTERVENTIONS:
Drug: 5% simvastatin ointment — 5% simvastatin ointment will be applied directly on IH lesion twice per day for 24 weeks

SUMMARY:
This is a 24-week, open-label pilot study to evaluate the safety and preliminary efficacy of 5% simvastatin ointment in treating 12 children with superficial IH.

The primary objective:

To evaluate the safety and tolerability of topical treatment with 5% simvastatin ointment for superficial IH over 24 weeks.

The secondary objective:

1.1 To evaluate the efficacy of 5% simvastatin ointment when topical treatment is administered twice daily for 24 weeks. Evaluation is performed at each clinic visit via investigator global assessment (IGA) based on standardized 3D digital photography and hemangioma activity score (HAS).

1.2 To evaluate the impact of 5% simvastatin ointment on quality of life using the IH-QoL questionnaire.

ELIGIBILITY:
Inclusion Criteria:

* Healthy children aged between 3 months and 5 years.
* Newly diagnosed superficial IH or experiencing rebound growth with a superficial component.
* Participants must possess at least one IH lesion with the longest diameter equal to or greater than 2 cm, located on any part of the body except the lips.
* Participants must not have received any of the following treatments for their IH:

  * Topical medical therapy within the past 2 weeks.
  * Systemic medical therapy within the past 3 months.
  * Laser treatment within the past 6 weeks.
* Written informed consent from the parent(s)/guardian(s) of minor participants must be obtained before any study procedure is performed.

Exclusion Criteria:

* IH is primarily characterized as subcutaneous, and deep, with minimal cutaneous involvement for evaluation.
* IH with active ulceration.
* IH to be treated involving the lips mainly.
* Participants with concurrent skin conditions that may impede accurate clinical assessment of the IH.
* Participants with hereditary or metabolic disorders requiring systemic statin therapy.
* Participants who are allergic to statins, or other ingredients present in the topical medication.

Ages: 3 Months to 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 12 (Estimated)
Dates: Start 2024-04-01 (Estimated); Primary Completion 2025-07-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Number of Participants with Treatment-Related Adverse Events | Baseline through week 24

SECONDARY OUTCOMES:
Percentage of participants achieved a 50% HAS reduction at week 12 compared to baseline | Baseline through week 12
Percentage of participants achieved a 75% HAS reduction from baseline by the end of the study (week 24) compared to baseline. | Baseline through week 24
Percentage of targeted hemangiomas with complete or nearly complete resolution (IGA 0 or 1), defined as a minimal degree of telangiectasia, skin thickening, and no definitive palpable cutaneous texture changes. | Baseline through week 24
Percentage of targeted hemangiomas that are stabilized (no noticeable change to baseline) or continue to progress. | Baseline through week 24
Percentage of participants with a significant improvement in quality-of-life, defined as > 50% reduction in the IH-QoL questionnaire score from baseline to week 24. | Baseline through week 24

CONTACTS AND LOCATIONS:
Overall Officials: Joyce Teng, MD, PhD, Principal Investigator — Stanford University
Locations (1):
- Stanford University, Palo Alto, California, United States

IPD SHARING:
Plan to Share IPD: No